CLINICAL TRIAL: NCT01043133
Title: Social Marketing in Medical Education: Influencing Medical Student Use of Evidence-based Templates in Outpatient Documentation of Asthma Care Using an Electronic Medical Record
Brief Title: Study of Medical Student Use of Templates to Document Outpatient Asthma Care in Electronic Medical Record
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Uniformed Services University of the Health Sciences (U.S. Federal Agency)
Responsible Party: Ronald W. Gimbel, PhD, Uniformed Services University of the Health Sciences
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Health Services Research
Other Study IDs: B02930
Record Dates: First submitted 2010-01-05; First posted 2010-01-06 (Estimated); Results first posted 2011-08-12 (Estimated); Last update posted 2011-08-12 (Estimated); Status verified 2010-01

CONDITIONS: Disease
Keywords: electronic medical records; documentation templates; clinical encounter notes
MeSH Terms: conditions — Disease

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No

ARMS (2):
- Intervention group (Experimental)
  Interventions: Behavioral: social marketing-based medical education intervention
- Control Group (No Intervention)

INTERVENTIONS:
Behavioral: social marketing-based medical education intervention — social-marketing based medical education intervention designed to influence medical student use of evidence-based templates. Led by physician instructor.
  Other Names: persuasion
  Arms: Intervention group

SUMMARY:
The purpose of the study is to measure the effectiveness of a social marketing-based medical education intervention on student use of evidence-based templates for documenting outpatient asthma care within an electronic medical record.

DETAILED DESCRIPTION:
The purpose of the study was to measure the effectiveness of a physician-educator led clinical documentation workshop, embedded with 7 persuasive social-marketing based messages, on medical student response using a targeted asthma template. Stated differently, whether a physician-educator could "persuade" medical students to use an evidence-based EMR asthma template to document an outpatient mild persistent asthma encounter with a patient.

ELIGIBILITY:
Inclusion Criteria:

* Third year medical student completing family medicine clerkship Uniformed Services University

Exclusion Criteria:

* All students other than those listed above

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 155 (Actual)
Dates: Start 2009-07; Primary Completion 2010-06 (Actual); Study Completion 2010-06 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Mark B. Stephens, MD, MS, Study Director — Uniformed Services University of the Health Sciences

RESULTS

PARTICIPANT FLOW:
Recruitment Details: All 3rd year USU medical students rotating through Family Medicine clerkship were invited to participate. The clerkship groups scheduled every 6-8 weeks during the 2009/10 academic year. The study included both male and female participants; ratio based on assignment to rotation group which is predetermined by medical school administrative staff.
Groups:
- Intervention Group: Students exposed to educational workshop on clinical documentation that was embedded with 7 select social marketing-based persuasion messages; reenforced behavior-seeking and behavior-avoidance based on template use.
- Control Group: Students exposed to clinical documentation workshop void of any of the 7 social marketing-based persuasion messages included in the intervention.
Period: Overall Study
Arm/Group | Intervention Group | Control Group
Started | 75 | 80
Completed | 74 | 78
Not Completed | 1 | 2

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Intervention Group | Control Group | Total
Number analyzed (Participants) | 75 | 80 | 155
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 75 | 80 | 155
  >=65 years | 0 | 0 | 0
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 26 | 33 | 59
  Male | 49 | 47 | 96
Region of Enrollment [Number; unit: participants]
  United States | 75 | 80 | 155

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants Using Evidence-based Template to Document Asthma Care Within an Electronic Medical Record
Description: The primary outcome measure is a count of whether or not the research participant uses the electronic health record-based Asthma AIM form to document a simulated outpatient mild persistent asthma encounter at T1 (immediately following intervention) and T2 (upon completion of family medicine clerkship approximately 35 days later).
Time Frame: immediately after invervention and 30+ days in follow-up
Measure: Number; unit: participants
Arm/Group | Intervention Group | Control Group
Number analyzed (Participants) | 75 | 80
participants | 41 | 11
Statistical Analysis 1: Comparison: Intervention Group vs Control Group; Test type: Superiority or Other; p = .01, log-binomial regression; log-binomial = 3.97, 95% CI 2-sided [1.34 to 11.79], Standard Error of Mean 3.97 — Robust Huber-White standard errors account for clustering

2. Secondary Outcome: Clinical Note Completeness Score
Description: The Note Completeness Score is a total score (range 1-31)earned when a clinical encounter note is compared against a note completeness score assessment tool designed by our research team. The tool measures 11 documentation components of the outpatient note. Each of the 11 components are scaled either 0-1 or 0-4 based on perceived importance by our physician designers.
Time Frame: immediately after intervention and 30+ days in follow-up
Measure: Mean (Standard Deviation); unit: score
Arm/Group | Intervention Group | Control Group
Number analyzed (Participants) | 75 | 80
score | 16.04 (2.78) | 17.05 (2.58)
Statistical Analysis 1: Comparison: Intervention Group vs Control Group; Test type: Superiority or Other; p = .05, ANCOVA; Mean Difference (Final Values) = -1.25, 95% CI 2-sided [-2.48 to -.03], Standard Deviation 2.78

ADVERSE EVENTS:
Arm/Group | Intervention Group | Control Group
Serious Adverse Events (participants affected / at risk) | 0/75 | 0/80
Other Adverse Events (participants affected / at risk) | 0/75 | 0/80

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes